CLINICAL TRIAL: NCT03122028
Title: A Prospective, Non-Randomized, Multi-Center, Open-Label, Non-Comparative, Interventional Clinical Investigation of the LAmbre Left Atrial Appendage Closure System
Brief Title: Clinical Investigation of the LAmbre Left Atrial Appendage Closure System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA-EU-01
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: LAmbre
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LAmbre closure system (Experimental)
  Interventions: Device: LAA closure system

INTERVENTIONS:
Device: LAA closure system — Patients with non-valvular paroxymal, persistent or permanent atrial fibrillation with long-term sustainability and cannot be treated with anticoagulation and scheduled for interventional left atrial appendage closure.

SUMMARY:
The aim of the study LA-EU-01 was to examine the safety and the feasibility of the LAmbreTM Left Atrial Appendage Closure System in patients with non-valvular paroxymal, persistent or permanent atrial fibrillation, by using imaging approaches, i.e. combined trans-esophageal and transthoracic echocardiography.

The conducted LA-EU-01 study was a prospective, non-randomized, multi-center, open-label, non-comparative, interventional clinical investigation with the participation of two clinical centers in Germany and the inclusion of 61 subjects.

Participating subjects were patients with non-valvular paroxymal, persistent or permanent atrial fibrillation with long-term sustainability and scheduled for interventional closure of the left atrial appendage who could not be treated with anticoagulation.

After the procedure of implantation of the LAmbreTM Left Atrial Appendage Closure System, patients underwent a first follow up assessment prior to hospital discharge then at 30 days, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients scheduled for interventional closure of the left atrial appendage (LAA) due to a high thromboembolic risk and cannot be treated with anticoagulation.
* Chronic atrial fibrillation ≥3 months; paroxysmal, persistent or permanent nonvalvular Atrial Fibrilation (AF)
* CHA2DS2 -VASC score 2 or higher
* Eligible for clopidogrel and aspirin
* Able to understand the requirements of the study and willing to follow study instructions, provide written informed consent, and agree to comply with all study requirements, including the required study follow-up visits

Exclusion Criteria:

* Presence of rheumatic, degenerative or congenital valvular heart diseases
* Presence of rheumatic, degenerative or congenital valvular heart diseases
* The diameter of left atrium ≥65 mm
* LAA Ostium < 12mm or > 30 mm
* Prior surgical removal of Left atrium
* Prior heart transplant
* Symptomatic patients with carotid artery disease (such as carotid stenosis ≥ 50%)
* Recent or acute myocardial infarction (MI) or unstable angina (recent is defined as within 3 months of implant date)
* Decompensated heart failure (NYHA grade III-IV)
* Patients have an electrophysiological ablation procedure planned within 30 days of potential the LAmbreTM Left Atrial Appendage Closure System implant date
* Patients have a planned electrophysiologic 30 days post implantation of the LAmbreTM Left Atrial Appendage Closure System
* Patients have a planned cardioversion 30 days post implantation of the LAmbreTM Left Atrial Appendage Closure System
* Patients with a history of heart valve replacement operation with an mechanical prosthesis
* History of stroke or Transient Ischemic Attack (TIA) within 30 days
* Have thrombocytopenia (platelet ≤ 100.000 platelets per microliter (mcL))
* Heart rate in rest > 110 beats per minute (BPM)
* A single episode of transient atrial fibrillation
* Pericardial effusion > 5mm pre-procedural
* Presence of active sepsis or endocarditis
* Cardiac tumors or other malignancy with estimated life expectancy less than 2 years
* Patients who are pregnant, breastfeeding, or desires to become pregnant during the course of the study
* Participation in the other investigational trials in which the primary endpoint is not met yet
* Subject dependency of the Sponsor, of the institution in which the trail is conducted, or of the investigator
* Investigator expectation that the patient will not be able to complete the trial according to the requirements
* A known allergy to nitinol Esophageal ultrasonic exclusion criteria
* LVEF ≤ 30 %
* Presence of thrombus in the left atrial appendage (LAA)
* Patent Foramen Ovale (PFO) with history of paradoxical embolism
* Mitral valve stenosis (Mitral valve area ≤ 2 cm2)
* Presence of complex aortic plaque (≥4mm) in ascending aorta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2016-03-09 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Serious adverse events | 6 months
  Absence of device or procedure related serious adverse events at 6 months after device implantation
Stable device placement | 6 months
  Stable device placement in left atrial appendage as assessed by transesophageal echocardiogram (TEE) at 6 months after device implant
Residual jet flow | 6 months
  Successful sealing around the device at the LAA orifice (residual jet flow of < 5 mm) as measured by transesophageal echocardiogram (TEE) at 6 months after device implant

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, Principal Investigator — The Cardiovascular Center